CLINICAL TRIAL: NCT06629207
Title: Artificial Intelligence on Molecular Imaging to Predict the Risks of Parkinson's Disease for Patients With Rapid Eye Movement Sleep Behavior Disorder
Brief Title: Artificial Intelligence in Molecular Imaging: Predicting Parkinson's Risk in REM Sleep Behavior Disorder
Acronym: NUK-RBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-00816
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder; Dementia, Lewy Body
Keywords: Parkinson Disease; Artificial Intelligence; REM Sleep Behavior Disorder
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder; Lewy Body Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NUK-RB Study (Experimental)
  Interventions: Device: PET/CT with 18-FDG; Device: SPECT : 123 I-FP-CIT (DATSCAN); Device: MRI

INTERVENTIONS:
Device: PET/CT with 18-FDG — FDG-PET scans will be acquired in a Siemens Biograph Vision Quadra PET/CT (Siemens, Germany) at 30-minute post-injection of approximately 80 MBq 18F-FDG. The duration of the acquisition is 20 minutes. The PET images will be reconstructed with the vendor's time of flight (TOF) point-spread-function (PSF) algorithm, following corrections for randoms, scatter, and decay. Attenuation correction will be performed first using low-dose CT.
Device: SPECT : 123 I-FP-CIT (DATSCAN) — DaT-Scans will be acquired in a GE Discovery NM/CT 670 Pro™. After injection of approximately 110 MBq 123I-FP-CIT, images will be acquired within 4 h post-injection. The duration of the acquisition is 35 minutes.
Device: MRI — MRI examination to exclude structural brain anomalies.

SUMMARY:
The study aims to systematically document the course of REM sleep behavior disorder (RBD) and investigate possible clinical and imaging biomarkers for disease progression and conversion risk to Parkinson's disease (PD), dementia with Lewy bodies (DLB), and multiple system atrophy (MSA). The study will use artificial intelligence to analyze imaging and develop a reliable method to predict and stratify patients approaching conversion to overt a-synucleinopathy. Participants will be clinically evaluated and 2 imaging procedures will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed clinical iRBD diagnosis by movement disorder specialists according to the International Classification of Sleep Disorders
2. Written informed consent

Exclusion Criteria:

1. Known diagnosis of PD or other neurodegenerative disorder
2. Unequivocal signs of parkinsonism on examination
3. Narcolepsy or other known causes of RBD
4. Moderate to severe obstructive sleep apnea
5. Abnormal neurological or MRI examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Deep Learning Model Accuracy in Predicting Neurodegenerative Conversion in isolated REM sleep behavior disorder (iRBD) through Early Biomarker Detection | From enrollment to end of follow-up period, expected to be 48 months
  The investigators aim to evaluate the predictive accuracy of a deep learning model in identifying patients with iRBD who will progress to a neurodegenerative disorder. The primary outcome will assess the model's sensitivity in detecting early imaging biomarkers linked to disease progression, with the goal of enabling earlier intervention and improving long-term outcomes.

SECONDARY OUTCOMES:
Comparison of the Estimated versus Observed Annual Conversion Risk of Isolated Rapid Eye Movement Behavior Disorder (iRBD) to Neurodegenerative Disorders | From enrollment to end of follow-up period, expected to be 48 months
  The investigators aim to compare the estimated annual conversion risk of 6.3% in patients with iRBD to Parkinson's disease or another overt alpha-synucleinopathy with the conversion rates observed in the study.
Evaluation of Deep Learning Model Accuracy in Predicting Conversion of Isolated REM Sleep Behavior Disorder (iRBD) to Parkinson's Disease | From enrollment to end of follow-up period, expected to be 48 months
  The investigators aim to evaluate the accuracy, receiver operating characteristic curves and area under the curve, specificity, and positive and negative predictive values of the applied deep learning method, predicting the conversion risk from iRBD to Parkinson's disease or another overt alpha-synucleinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Kuanggyu Shi, Prof. Dr. ing., Principal Investigator — University Bern, Inselspital, Center for Artificial Intelligence in Medicine
Locations (1):
- Inselspital, University Clinic for Nuclear Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No